CLINICAL TRIAL: NCT04814056
Title: An Open-Labeled, Single-Arm Clinical Study to Evaluate the Efficacy of Afatinib in Treatment of Locally Advanced or Metastatic Non-Small Cell Lung Cancer With NRG1-Fusion
Brief Title: To Evaluate the Efficacy of Afatinib in the Treatment of Locally Advanced/Metastatic Non-Small Cell Lung Cancer With NRG1 Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Lu Shun, Chief physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BI-IIT-AFATINIB-I
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: NRG1-fused Non-small Cell Lung Cancer
Keywords: Locally advanced (stage IIIB) or metastatic (stage IV); have previously received platinum-based doublet chemotherapy and developed disease progression subsequently
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Afatinib treatment group (Experimental): This is an open-label, sing-arm phase IV clinical study
  Interventions: Drug: Afatinib Dimaleate

INTERVENTIONS:
Drug: Afatinib Dimaleate — Afatinib is the second-generation TKI drug, which can irreversibly bind to receptors of erbB family. Afatinib will be administered orally at a dose of 40 mg per time, Q.D. If a patient cannot tolerate a dose of 40mg due to adverse reactions, when the adverse reactions restore to level 1 (CTCAE 5.0) or below, the dosage could be adjusted to 30mg per day, Q.D.
  Other Names: GIOTRIF®

SUMMARY:
This is an open-label, sing-arm, phase IV clinical study. The study is designed to evaluate the efficacy of Afatinib in treatment of NRG1-fused locally advanced/metastatic non-small cell lung cancer (NSCLC), and explore the clinical factors that may predict the effectiveness of treatment.

DETAILED DESCRIPTION:
This is an open-label, sing-arm clinical study,which will recruit about 15 patients in China.

The study is designed to evaluate the efficacy of Afatinib in treatment of NRG1-fused locally advanced/metastatic non-small cell lung cancer (NSCLC), and explore the clinical factors that may predict the effectiveness of treatment.

Target Patient Population:Locally advanced (stage IIIB) or metastatic (stage IV) NRG1-fused non-small cell lung cancer patients, who have previously received platinum-based doublet chemotherapy and developed disease progression subsequently.

Test Drug, Dosage and Medication Regimen:Afatinib is the second-generation TKI drug, which can irreversibly bind to receptors of erbB family. Afatinib will be administered orally at a dose of 40 mg per time, Q.D. If a patient cannot tolerate a dose of 40mg due to adverse reactions, when the adverse reactions restore to level 1 (CTCAE 5.0) or below, the dosage could be adjusted to 30mg per day, Q.D.

Evaluations of Study:The data to be collected include demographic characteristics of the patients, information necessary to determine whether the patients are qualified (including medical history, features of previous and current diseases and NRG1 fusion status in tumor tissue), and efficacy and safety data in terms of objective response rate (ORR), disease control rate (DCR) and progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* The patient or his/her legal representative has signed a written informed consent form and dated it prior to any specific research procedure.
* Aged 18 years or older.
* Locally advanced or metastatic non-small cell lung cancer with NRG1 fusion detected by DNA or RNA-based next-generation sequencing (NGS) technology in tumor tissue specimens or liquid specimens.
* The patient has received platinum-based doublet chemotherapy previously.
* ECOG performance status score is 0~2.
* The patient has sufficient bone marrow and organ functionality, which can be proved by complete blood cell count, blood biochemistry and urine biochemistry tests at baseline.
* The patient has measurable lesion(s).
* The female patient of childbearing age must adopt appropriate contraceptive measures and are not allowed to breastfeed a child.
* The male patient must voluntarily use contraceptives.

Exclusion Criteria:

* The patient has shown any severe or uncontrollable systemic disease sign that the investigators believe may significantly change the risk/benefit balance of the patient, including uncontrollable hypertension, high active bleeding tendency, active infection or significant damage of bone marrow or other functions.
* The patient has previously been treated with EGFR-TKI or any monoclonal antibody that acts on HER2/3.
* The patient has been found with symptomatic metastatic tumor of central nervous system (CNS).
* The patient has a history of interstitial pneumonia or radiation pneumonia requiring steroid therapy.
* The patient has not recovered yet from toxic reactions with CTCAE grade ≥3 (CTCAE5.0) caused by previous treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-09-29 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | Up to 12 months
  ORR

SECONDARY OUTCOMES:
disease control rate (DCR) | Up to 12 months
  DCR
progression-free survival (PFS) | Up to 12 months
  PFS

CONTACTS AND LOCATIONS:
Overall Officials: Yongfeng Yu, Master, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No